CLINICAL TRIAL: NCT06265454
Title: Effect of Low Concentration Atropine Eye Drops on Choroidal Thickness, Central Corneal Thickness, Anterior Scleral Thickness and Axial Length in Myopic Children
Brief Title: Low Dose Atropine Eye Drops in Myopic Egyptian Children
Acronym: LAMP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, aya mahmoud, Doctor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LDAED IN MC
Record Dates: First submitted 2024-02-11; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Myopia Progression; Axial Length, Eye; Sclera Thickness
Keywords: myopia; low dose; atropine eye drops; mypoic children; myopia progression; LAMP
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- myopic children atropine 0.05% (Active Comparator): they will receive topical atropine 0.05% for 12 weeks and all investigations will be done before administration of atropine (baseline assessment), then after 1 month, 2 months, 3 months.
  Interventions: Drug: low dose atropine eye drops
- myopic children atropine 0.01% (Active Comparator): they will receive topical atropine 0.01% for 12 weeks and all investigations will be done before administration of atropine (baseline assessment), then after 1 month, 2 months, 3 months.
  Interventions: Drug: low dose atropine eye drops
- myopic children placebo (Placebo Comparator): they will receive placebo for 12 weeks and all investigations will be done before administration of placebo (baseline assessment), then after 1 month, 2 months, 3 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: low dose atropine eye drops — Atropine is a nonselective muscarinic antagonist used for myopia control in previous studies.
  Arms: myopic children atropine 0.01%; myopic children atropine 0.05%
Drug: Placebo — placebo
  Arms: myopic children placebo

SUMMARY:
Previous Studies reported that low concentration atropine eye drops may be effective in increasing the choroidal blood flow and thickness and this slows myopia progression.

purpose of the study is to compare changes in axial length, anterior chamber depth, choroidal thickness, central corneal thickness and anterior scleral thickness among myopic children receiving atropine 0.05% or 0.01% and placebo.

DETAILED DESCRIPTION:
Myopia is the most common refractive error, and its prevalence rate is increasing worldwide, as per WHO, it is projected to increase from 22% in 2000 to 52% by 2050. It is more prevalent in developed, industrial areas and affects individuals of all ages (Singh et al., 2022). Myopia, especially the degenerative type, is associated with sight-threatening complications, including presenile cataract, glaucoma, retinal detachment, choroidal neovascularization, myopic macular degeneration, scleral and choroidal thinning (Sanchez-Cano et al., 2014 and Gupta et al., 2015) which makes myopia a major public health concern and finding an effective treatment to prevent myopia progression is critical (Wakazono et al., 2016).

Atropine is a nonselective muscarinic antagonist used for myopia control in previous studies. However, its actual mechanism of action is not well known (Yam et al., 2019).

But different mechanisms were described, first mechanism, that atropine may induce release of dopamine causing thickening of choroid (Nickla et al., 2010) Second mechanism,blockage of choroidal smooth muscle contraction through its anti-muscarinic action. Third one, increasing capillary permeability. Fourth, potentiating the synthesis and release of intraocular nitric oxide (Yam et al.,2022) also it stimulates retinal expression of the transcription factor ZENK which was considered an eye growth-inhibiting signal (Torii et al., 2017). All these mechanisms cause thickening of the choroid and increased choroidal blood flow which has been found to play a role in the regulation of eye growth and refractive error development through inhibition of the penetration of various retinal-derived growth factors that act as mechanical barriers and slow scleral growth (Nickla et al., 2015 & Guggenheim et al., 2011). Also, choroid can secrete growth factors that prevent scleral hypoxia (Wu et al., 2018).

According to the Low-concentration Atropine for Myopia Progression (LAMP) study, different atropine eye drops concentrations 0.05%, 0.025%, and 0.01% controlled myopia progression but the most effective concentration on spherical equivalent and axial length progression was 0.05% (Yam et al., 2019).

Zhang et al. reported in 2016 that administration of 1% atropine gel increased the choroidal thickness in young Chinese children with inhibition of eye growth.

Also, jiang et al. in 2021 mentioned that after one week of administration of 1% atropine significant changes in spherical equivalent, axial length and choroidal thickness and after cessation of the medication for 7 weeks those returned to baseline levels.

In 2022, Zhou et al. reported also increased sub foveal choroidal thickness and in all quadrants in myopes in contrast to increased thickness in nasal quadrant only in hyperopes and non-significant change in emmetropes.

A recent study in 2023 found a dose dependent ocular biometrics changes, including axial length and anterior chamber depth, during low-dose atropine treatment in children with myopia (Hvid-Hansen et al., 2023).

In Li et al. study in 2021 they mentioned that younger children required higher atropine concentrations to show better responses.

In 2023, Zhou et al. reported thinner anterior sclera in myopes compared to emmetropes and a negative correlation between anterior scleral thickness (AST)and axial length and recommended usage of AST as a tool for monitoring of myopia progression.

Optical Coherence Tomography (OCT) is a non-invasive imaging modality, it was first reported in 1991 as a diagnostic technology that provides a cross-sectional image of the retina and choroid. It creates a cross-sectional map of the retina based on low-coherence interferometry (Aumann et al., 2019).

There are two types of OCT, time domain OCT and spectral domain OCT but the most widely used now is spectral domain OCT as it has scan rate between 20,000 and 40,000 per second which improves resolution and reduces the likelihood of missing lesions (Xie et al., 2021).

ELIGIBILITY:
Inclusion Criteria:

* Age ranges from 6 to 12.
* Spherical equivalent ≥ -1.0 D.

Exclusion Criteria:

* Astigmatism ≥ 3.0 D.
* History of allergy to atropine or positive skin allergy test.
* Ocular pathology otherwise myopia.
* Recent ocular surgery.
* Chronic systemic disease.
* Use of rigid contact lenses or soft contact lenses for 1 week before participating in the study

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
change in the average Choroidal Thickness over follow up period. | from enrollment till end of eye drops trial over 3 months and after stopping the drops for 3 months
  Follow up of choroidal thickness during treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Aya Mahmoud, Master's, Principal Investigator — Ain Shams University
Locations (1):
- Ain shams university, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Z, Zhou Y, Xie Z, Chen T, Gu Y, Lu S, Wu Z. The effect of topical atropine on the choroidal thickness of healthy children. Sci Rep. 2016 Oct 7;6:34936. doi: 10.1038/srep34936. PMID 27713535
- [Background] Zhou J, He H, Yang Q, Wang JY, You ZP, Liu LL. Comparison of anterior sclera thickness in emmetropes and myopes. BMC Ophthalmol. 2023 Feb 14;23(1):67. doi: 10.1186/s12886-023-02775-x. PMID 36782174
- [Background] Ye L, Shi Y, Yin Y, Li S, He J, Zhu J, Xu X. Effects of Atropine Treatment on Choroidal Thickness in Myopic Children. Invest Ophthalmol Vis Sci. 2020 Dec 1;61(14):15. doi: 10.1167/iovs.61.14.15. PMID 33320168
- [Background] Yam JC, Jiang Y, Tang SM, Law AKP, Chan JJ, Wong E, Ko ST, Young AL, Tham CC, Chen LJ, Pang CP. Low-Concentration Atropine for Myopia Progression (LAMP) Study: A Randomized, Double-Blinded, Placebo-Controlled Trial of 0.05%, 0.025%, and 0.01% Atropine Eye Drops in Myopia Control. Ophthalmology. 2019 Jan;126(1):113-124. doi: 10.1016/j.ophtha.2018.05.029. Epub 2018 Jul 6. PMID 30514630
- [Background] Xie R, Qiu B, Chhablani J, Zhang X. Evaluation of Choroidal Thickness Using Optical Coherent Tomography: A Review. Front Med (Lausanne). 2021 Dec 3;8:783519. doi: 10.3389/fmed.2021.783519. eCollection 2021. PMID 34926529
- [Background] Wang Y, Zhu X, Xuan Y, Wang M, Zhou X, Qu X. Short-Term Effects of Atropine 0.01% on the Structure and Vasculature of the Choroid and Retina in Myopic Chinese Children. Ophthalmol Ther. 2022 Apr;11(2):833-856. doi: 10.1007/s40123-022-00476-0. Epub 2022 Feb 20. PMID 35184254
- [Background] Wakazono T, Yamashiro K, Miyake M, Nakanishi H, Oishi A, Ooto S, Tsujikawa A, Yoshimura N. Association between Eye Shape and Myopic Traction Maculopathy in High Myopia. Ophthalmology. 2016 Apr;123(4):919-21. doi: 10.1016/j.ophtha.2015.10.031. Epub 2015 Dec 11. No abstract available. PMID 26686963
- [Background] Torii H, Ohnuma K, Kurihara T, Tsubota K, Negishi K. Violet Light Transmission is Related to Myopia Progression in Adult High Myopia. Sci Rep. 2017 Nov 6;7(1):14523. doi: 10.1038/s41598-017-09388-7. PMID 29109514
- [Background] Singh H, Singh H, Latief U, Tung GK, Shahtaghi NR, Sahajpal NS, Kaur I, Jain SK. Myopia, its prevalence, current therapeutic strategy and recent developments: A Review. Indian J Ophthalmol. 2022 Aug;70(8):2788-2799. doi: 10.4103/ijo.IJO_2415_21. PMID 35918918
- [Background] Sanchez-Cano A, Orduna E, Segura F, Lopez C, Cuenca N, Abecia E, Pinilla I. Choroidal thickness and volume in healthy young white adults and the relationships between them and axial length, ammetropy and sex. Am J Ophthalmol. 2014 Sep;158(3):574-83.e1. doi: 10.1016/j.ajo.2014.05.035. Epub 2014 Jun 5. PMID 24907431
- [Background] Nickla DL, Totonelly K, Dhillon B. Dopaminergic agonists that result in ocular growth inhibition also elicit transient increases in choroidal thickness in chicks. Exp Eye Res. 2010 Nov;91(5):715-20. doi: 10.1016/j.exer.2010.08.021. Epub 2010 Aug 27. PMID 20801115
- [Background] Nickla DL, Totonelly K. Choroidal thickness predicts ocular growth in normal chicks but not in eyes with experimentally altered growth. Clin Exp Optom. 2015 Nov;98(6):564-70. doi: 10.1111/cxo.12317. PMID 26769180
- [Background] Jiang Y, Zhang Z, Wu Z, Sun S, Fu Y, Ke B. Change and Recovery of Choroid Thickness after Short-term Application of 1% Atropine Gel and Its Influencing Factors in 6-7-year-old Children. Curr Eye Res. 2021 Aug;46(8):1171-1177. doi: 10.1080/02713683.2020.1863431. Epub 2021 Jan 4. PMID 33390025
- [Background] Hvid-Hansen A, Jacobsen N, Hjortdal J, Moller F, Ozenne B, Kessel L. Low-Dose Atropine Induces Changes in Ocular Biometrics in Myopic Children: Exploring Temporal Changes by Linear Mixed Models and Contribution to Treatment Effect by Mediation Analyses. J Clin Med. 2023 Feb 17;12(4):1605. doi: 10.3390/jcm12041605. PMID 36836139
- [Background] Gupta P, Jing T, Marziliano P, Cheung CY, Baskaran M, Lamoureux EL, Wong TY, Cheung CM, Cheng CY. Distribution and determinants of choroidal thickness and volume using automated segmentation software in a population-based study. Am J Ophthalmol. 2015 Feb;159(2):293-301.e3. doi: 10.1016/j.ajo.2014.10.034. Epub 2014 Nov 5. PMID 25447120
- [Background] Guggenheim JA, Chen YP, Yip E, Hayet H, Druel V, Wang L, Erichsen JT, Tumlinson AR, Povazay B, Drexler W, Hocking PM. Pre-treatment choroidal thickness is not predictive of susceptibility to form-deprivation myopia in chickens. Ophthalmic Physiol Opt. 2011 Sep;31(5):516-28. doi: 10.1111/j.1475-1313.2011.00827.x. Epub 2011 Mar 29. PMID 21446921
- See also: 10.1159/000526448 — https://pubmed.ncbi.nlm.nih.gov